CLINICAL TRIAL: NCT02158702
Title: Prospective Follow-up of Relapse Myeloma Patients After Previous Exposure to Bortezomib and Lenalidomide Treated on Pomalidomide and Dexamethasone
Brief Title: Efficacy and Toxicity Study of Pomalidomide and Dexamethasone in Patients Who Have Relapsed After Exposure to Lenalidomide and Bortezomib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Haematology-Oncology, Senior Consultant, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00498
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma; Relapse After Use of Lenalidomide and Bortezomib
Keywords: Relapsed Myeloma Patients; Relapsed after use of Bortezomib and Lenalidomide; Pomalidomide and Dexamethasone; Efficacy and Safety
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide and Dexamethasone (Experimental): PO pomalidomide 4mg from D1-21 and PO dexamethasone 40mg D1, 8, 15 and 22 in a 28-day cycle.
  PO or IV cyclophosphamide 300mg/m2 on D1, 8 and 15 can be added at the discretion of the treating physician to induce added response under the following circumstances: 1) If there is less than a MR after 3 cycles in the absence of disease progression, or 2) If there is disease progression within the first 3 cycles of Pomalidomide and Dexamethasone treatment.
  Patients will be assessed every 28 days (+/-10 days). Patients shall receive the treatment until disease progression, unacceptable toxicity as determined by treating physician, withdrawal of consent or mortality (whichever occurs first).
  Interventions: Drug: Pomalidomide and Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide and Dexamethasone — Pomalidomide will be given at 4mg once daily for 21 days in a 28-day cycle. Dexamethasone will be given at a dose of 40mg orally once a week for 4 weeks (D1,8,15,22).

SUMMARY:
Asian patients with relapsed myeloma after prior treatment with bortezomib and lenalidomide will treatment on pomalidomde and dexamethasone.

Baseline, follow-up, survival and toxicity information will be collected.

DETAILED DESCRIPTION:
Myeloma patients who relapse after prior treatment with bortezomib and lenalidomide have survival of less than 1 year. Recently, a randomized study of Pomalidomide and dexamethasone conducted in compared with placebo and dexamethasone showed that pomalidomide can improve survival of this group of patients.

Pomalidomide is a new immunomodulatory drug which has been shown to be active in myeloma patients who relapse after bortezomib and lenalidomide. A recent phase III study comparing pomalidomide plus dexamethasone with placebo plus high dose dexamethasone in patients with prior exposure to bortezomib and lenalidomide, showed that the use of pomalidomide significantly improve the overall survival of these patients. However, this study did not include Asian patients. Therefore the efficacy and toxicity of pomalidomide remains to be described in Asian patients

ELIGIBILITY:
1. Multiple myeloma, diagnosed according to standard criteria, with relapsing and refractory disease at study entry
2. Patients must have evaluable multiple myeloma with at least one of the following (within 21 days of starting treatment)

   1. Serum M-protein ≥ 0.5g/dL, or
   2. In subjects without detectable serum M-protein, Urine M-protein ≥ 200mg/24 hour, or serum free light chai (sFLC) > 100mg/L (involved light chain) and an abnormal kappa/Lambda ratio
3. Can receive up to 6 lines of prior treatment. (Induction therapy followed by stem cell transplantation and consolidation/maintenance therapy will be considered as one line of treatment)
4. Must have failed lenalidomide (based on 1 of the following criteria: a) Refractory to lenalidomide; or b) no better than stable disease after 3 cycles of lenalidomide) and relapsed from previous treatment with bortezomib. Refractoriness is defined as disease progression on treatment or progression within 6 months after the last dose of a given therapy. Relapse is defined according to the criteria of IMWG
5. Males and females ≥ 18 years of age or > country's legal age for adult consent
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
7. Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
   2. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   3. Calculated creatinine clearance ≥ 45mL/min or creatinine < 3mg/dL.
8. Female patients who:

   1. Are naturally postmenopausal for at least 2 year before enrolment
   2. Are surgically sterile
   3. If they are of childbearing potential**, agree to

      * adhere to the pomalidomide pregnancy prevention risk management program in Appendix 8 :
      * All women of childbearing potential must agree to have two negative pregnancy test within 10-14 days and 24hrs before commencing pomalidomide and use two reliable methods of contraception simultaneously or practice complete abstinence from any heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study; 2) while participating in the study; 3) dose interruptions; and 4) for at least 28 days after study treatment discontinuation. The two methods of reliable contraception must include one highly effective method and one additional effective method to prevent pregnancy, not plan on conceiving children during or within 6 months following pomalidomide. (See Appendix 8 Pregnancy Prevention and Risk Management Program)
9. Male patients, even if surgically sterilized (i.e. status post-vasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period and through 28 days after the last dose of study treatment, OR
   2. Agree to completely abstain from heterosexual intercourse, AND
   3. Must also adhere to the guidelines of the pomalidomide pregnancy prevention and risk management program
10. Written informed consent in accordance with federal, local and institutional guidelines

    * A female of childbearing potential (FCBP) is defined as a sexually mature woman who: 1 has not undergone a hysterectomy or bilateral oophorectomy or 2, has not been naturally post-menopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (I.E, has had menses at any time in the preceding 24 consecutive months).

1.1. Exclusion Criteria

1. Female patients who are lactating or pregnant
2. Multiple Myeloma of IgM subtype
3. Glucocorticoid therapy (prednisolone > 30mg/day or equivalent) within 14 days prior to informed consent obtained
4. POEMS syndrome
5. Plasma cell leukemia or circulating plasma cells ≥ 2 x 109/L
6. Waldenstrom's Macroglobulinaemia
7. Patients with known amyloidosis
8. Chemotherapy with approved or investigation anticancer therapeutics within 21 days prior to starting pomalidomide treatment
9. Focal radiation therapy within 7 days prior to start of pomalidomide. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to start of pomalidomide
10. Immunotherapy (excluding steroids) 21 days prior to start of pomalidomide
11. Major surgery (excluding kyphoplasty) within 28 days prior to start of pomalidomide
12. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained
13. Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
14. Patients with known cirrhosis
15. Second malignancy within the past 3 years except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Breast carcinoma in situ with full surgical resection
16. Patients with myelodysplastic syndrome
17. Patients with steroid or lenalidomide hypersensitivity
18. Prior treatment with pomalidomide
19. Ongoing graft-versus-host disease
20. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to starting pomalidomide treatment
21. Contraindication to any of the required concomitant drugs or supportive treatments
22. Any clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-02 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
To assess the progression free survival (PFS) for pomalidomide and dexamethasone in patients who have relapsed and are refractory to lenalidomide and have previously been treated with bortezomib | 2 year

SECONDARY OUTCOMES:
To assess Overall Response Rate (ORR) | 2 year
To see if addition of cyclophosphamide with induce additional response in patient who do not achieve an minimal response (MR) after 3 months | 2 year
To assess Overall Survival (OS) | 5 year
To assess Duration of Response (DOR) | 2 year
To assess Safety and Tolerability | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Wee Joo Chng, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore